CLINICAL TRIAL: NCT06019507
Title: A 60 Month, Single-arm, Proof-of-concept Study to Induce Allogeneic Tolerance in Deceased Donor Liver Transplant Recipients Using Siplizumab, an Anti-CD2 Antibody in Combination With Cyclophosphamide and Splenectomy
Brief Title: A Study of TCD601 in the Induction of Tolerance in de Novo Liver Transplantation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ITB-Med LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TCD601G201
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Liver Transplantation
MeSH Terms: interventions — siplizumab; Cyclophosphamide; Tacrolimus; Mycophenolic Acid; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): TCD601administered after liver transplant with splenectomy with cyclophosphamide and immunosuppression therapy
  Interventions: Biological: TCD601; Biological: Cyclophosphamide; Drug: TAC; Drug: MMF; Drug: Corticosteroids

INTERVENTIONS:
Biological: TCD601 — Investigational Product
  Other Names: siplizumab
Biological: Cyclophosphamide — Conditioning Regimen
Drug: TAC — Immunosuppression Therapy
  Other Names: Tacrolimus
Drug: MMF — Immunosuppression Therapy
  Other Names: Mycophenolate Mofetil
Drug: Corticosteroids — Immunosuppression Therapy

SUMMARY:
The purpose of this study is to evaluate if treatment with a siplizumab-based regimen can induce allogeneic tolerance in liver transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the study requirements and provide written informed consent before and study assessment is performed
* Adult subjects aged 18-70 receiving an ABO compatible deceased donor liver transplant
* Male study subjects willing to maintain barrier contraception (condom) and agree not to father a child until 12 weeks after the last dose of MMF

Exclusion Criteria:

* Pregnant or nursing (lactating) women
* Subjects with a history of TB or latent TB infection
* Subjects with a history of cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Number of Liver Transplant Recipients off of immunosuppression Therapy. | 30 months
  Determine if treatment with siplizumab can induce allogeneic tolerance in liver transplant recipients

SECONDARY OUTCOMES:
The Incidence of adverse events and serious adverse events | 30 months
  To explore the safety and tolerability of TCD601.

CONTACTS AND LOCATIONS:
Overall Officials: Kellie Kennon, BSN, Study Director — ITB-MED
Locations (1):
- Karolinska University Hospital, Stockholm, Huddinge, Sweden